CLINICAL TRIAL: NCT01981200
Title: Feasibility of Progressive Knee Extension Strength Training Using Ankle Weight Cuffs in Patients Hospitalized With COPD in Acute Exacerbation
Brief Title: Feasibility of Strength Training in Patients Hospitalized Due to COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederikssunds Hospital, Denmark (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Linette Marie Kofod, Physiotherapist, Frederikssunds Hospital, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210977
Record Dates: First submitted 2013-10-30; First posted 2013-11-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: COPD; Muscle Weakness
Keywords: COPD acute exacerbation; Physiotherapy; Resistance training; Muscle strength; Handheld dynamometer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscle Weakness | interventions — Resistance Training; Hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resistance training in AECOPD (Experimental): The patients conduct daily training during admission with weight cuff 3 set of 10 rep.
  Interventions: Other: Resistance training in AECOPD

INTERVENTIONS:
Other: Resistance training in AECOPD — The patients begin training on day 1 of admittance. The training consists of knee extension performed in the sitting position on the bed with a 90 degrees of flexion of the knees. The weight cuffs are tired to the angles with a weight corresponding to 10 RM (the weight lifted 10 times). The weights and exercises are subjected to supervision on daily basis by the physiotherapist. The weight is increased after every set of training if more than 10 rep. can be performed with a given weight. Limitations to exercise is also recorded along with the degree of dyspnoea as assessed by the Borg CR10, possible oxygen supplementation and saturation is recorded before and following exercise.
  Other Names: Weight cuffs; Strength training; hospitalization

SUMMARY:
To examine the feasibility of progressive unilateral knee-extension strength training using ankle weight cuffs in patients hospitalized due to acute exacerbation in COPD

DETAILED DESCRIPTION:
We decided that feasibility is indicated if: 1) the absolute training loads increase progressively, 2) more than 80% of the planned training sessions are completed, and 3)if the absolute training loads do not exceed 20 kg (2 x10kg weight cuffs) for 90% of patients.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of COPD
* Be admitted to the pulmonary ward due to an exacerbation in COPD
* Provide informed consent to participation in the study
* Be able to maintain an upright position on a chair
* Be able to be guided to training and understand instructions for participating

Exclusion Criteria:

Patients suffering from diseases that prevents the use of wrist weights such as

* Deep venous thrombosis (DVT)
* Erysipelas
* Painful edema of the limbs
* Lack of ability to walk, habitually
* Predicted hospital stay of less than four days as predicted by a pulmonary physician
* Patients admitted Friday night or Saturday morning cannot be stared up within 24 hours of admittance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Increase of training load during admission | The patients will be followed for the duration of hospital stay, an expected average of 6 days
  Change in training loads measured by the number of kilos lifted using ankle weight cuffs in 3 sets of 10 repetition maximum at the first training day to the number of kilos lifted at the last training day

SECONDARY OUTCOMES:
Maximal isometric knee extension strength | The patients will be followed for the duration of hospital stay, an expected average of 6 days
  Maximal isometric knee extension strength is measured unilaterally by a fixated handheld dynamometer. The test will be performed upon admission and at the day of discharge
Sit-to- stand- test | The patients will be followed for the duration of hospital stay, an expected average of 6 days
  The number of times the patient comes to full standing position in 30 seconds. The Sit to Stand test provides a measurement of a person's lower body (particularly quadriceps) strength. This is associated with the ability to perform lifestyle tasks such as climbing stairs, getting in and out of a vehicle or bath. The test will be performed upon admission and on the day of discharge
Timed Up and Go (TUG) | The patients will be followed for the duration of hospital stay, an expected average of 6 days
  A test used to assess a person's mobility and requires both static and dynamic balance. The time that a person takes to rise from a chair, walk three metres, turn around, walk back to the chair, and sit Down. The test will be performed at admission and at the day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Linette M Kofod, PT, Principal Investigator — Nordsjællands Hospital - Frederikssund; Morten T Kristensen, PhD, Study Chair — Copenhagen University Hospital, Hvidovre
Locations (1):
- Nordsjællands Hospital - Frederikssund, Frederikssund, Denmark